CLINICAL TRIAL: NCT02500615
Title: The Effect of Electronic Cigarette (ECIG) Liquid Vehicles on ECIG Acute Effects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HM20004850; 1F31DA040319-01 (NIH)
Record Dates: First submitted 2015-07-06; First posted 2015-07-16 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Nicotine Exposure; Nicotine Withdrawal Suppression

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (5):
- 0 PG: 100 VG (Experimental)
  Interventions: Other: ECIG liquid vehicles
- 30 PG: 70 VG (Experimental)
  Interventions: Other: ECIG liquid vehicles
- 50 PG: 50 VG (Experimental)
  Interventions: Other: ECIG liquid vehicles
- 70 PG: 30 VG (Experimental)
  Interventions: Other: ECIG liquid vehicles
- 100 PG: 0 VG (Experimental)
  Interventions: Other: ECIG liquid vehicles

INTERVENTIONS:
Other: ECIG liquid vehicles — The ratio of propylene glycol and vegetable glycerin will be changed while all other factors of the electronic cigarette provided to participants will be held constant.

SUMMARY:
This study examines the acute effects in ECIG users of the two primary vehicles in ECIG liquids, propylene glycol and vegetable glycerin. Thirty experienced ECIG users will use an ECIG in five conditions that will differ only by the propylene glycol:vegetable glycerin ratio: 100:0, 70:30, 50:50, 30:70, and 0:100 (device voltage, heater resistance, liquid nicotine concentration, puff number, and interpuff interval all will be held constant). Plasma nicotine concentration, subjective effects, and puffing behaviors will be recorded in each condition.

DETAILED DESCRIPTION:
Electronic cigarettes (ECIGs) are among the most important issues in public health today due to their dramatic increase in popularity. However, very little is known about ECIGs, including what factors may make them more likely to be used and abused. Examining factors that influence nicotine yield, delivery, and subjective effects from ECIGs is essential to understanding their abuse liability. Limited pre-clinical research has revealed that nicotine yield may be influenced by the ratio of the two liquid vehicles, propylene glycol (PG) and vegetable glycerin (VG), most commonly found in ECIG solutions. Specifically, higher proportions of PG result in greater nicotine yields. However, the influence of PG:VG ratio on nicotine delivery and subjective effects associated with ECIG use has not been examined previously. The primary hypotheses are that higher proportions of PG will result in greater nicotine delivery and subjective effect profiles suggestive of higher abuse liability in ECIG users. Results from this project will result in further understanding of the factors that influence the abuse liability of ECIGs and could inform regulation of these products.

ELIGIBILITY:
Inclusion Criteria:

* Participants must use ≥1 ml of ECIG solution daily
* Must use ECIG solution with a nicotine concentration ≥12 mg/ml
* Must have used an ECIG for ≥3 months
* Must be willing to abstain from nicotine and tobacco products for ≥12 hours prior to each session.

Exclusion Criteria:

* History of chronic disease or psychiatric condition
* Regular use of a prescription medication
* Marijuana use >10 and alcohol use >25 days in the past 30
* Any other illicit drug use (e.g., cocaine, opioids) in the past 30 days.
* Positive test for pregnancy (by urinalysis)
* Daily use of >5 conventional tobacco cigarettes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2016-07; Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Plasma nicotine concentration (ng/ml) | Collected at each of the 5 visits. Participants can complete up to 2 sessions/week. Thus the average time period to complete all 5 sessions is approximately 3 weeks. Each individual session is approximately 3 hours long.
  taken via intravenous catheter
Withdrawal suppression items on a visual analog scale | Collected at each of the 5 visits. Participants can complete up to 2 sessions/week. Thus the average time period to complete all 5 sessions is approximately 3 weeks. Each individual session is approximately 3 hours long.
  provided using computerized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tory R Spindle, B.S., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Clinical Behavioral Pharmacology Laboratory, Richmond, Virginia, United States